CLINICAL TRIAL: NCT05884554
Title: A PHASE 1, OPEN-LABEL, SINGLE-DOSE, PARALLEL GROUP STUDY TO ASSESS PHARMACOKINETICS, SAFETY AND TOLERABILITY OF PF-07817883 IN ADULT PARTICIPANTS WITH VARYING DEGREES OF HEPATIC IMPAIRMENT RELATIVE TO PARTICIPANTS WITHOUT HEPATIC IMPAIRMENT
Brief Title: A Study to Learn About How Loss of Liver Function Affects the Blood Levels of the Study Medicine Called PF-07817883.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: C5091014
Record Dates: First submitted 2023-05-23; First posted 2023-06-01 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: COVID-19
Keywords: Hepatic Impairment; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Experimental): No hepatic impairment
  Interventions: Drug: PF-07817883
- Cohort 2 (Experimental): Mild hepatic impairment
  Interventions: Drug: PF-07817883
- Cohort 3 (Experimental): Moderate hepatic impairment
  Interventions: Drug: PF-07817883
- Cohort 4 (Experimental): Severe hepatic impairment
  Interventions: Drug: PF-07817883

INTERVENTIONS:
Drug: PF-07817883 — Experimental

SUMMARY:
The purpose of the study is to learn about the safety of PF-07817883 and how PF-07817883 is processed in the body of adult participants. These participants will have different degrees of loss of liver function. Participants with mild, moderate, severe or no loss of liver function will be enrolled in 4 groups.

This study is seeking participants who:

* are male or female of 18- 75 years of age
* either have different amounts of damage to liver function or for one of the groups, no damage
* willing to follow the requirements of the study including stay at clinic for 6 nights and 7 days

About, 6-8 participants will be enrolled in group 1 (participants without loss of liver function) and group 3 (participants with moderate loss of liver function). In group 4 (participants with severe loss of function), around 4 to 8 participants will be enrolled. Participants in group 2 (mild loss of function) will only be enrolled after review of the data from groups 3 and 4.

If participants consent to participate in the study, it may take up to 4 weeks to complete all the tests to confirm if they are eligible to participate in the study. If they seem to be eligible for the study, participants will be admitted to a clinic research unit (CRU) at least 12 hours before dosing. On Day 1, participants will receive a single dose of study medicine (Day 1). A series of blood samples will be collected before and after dosing. Participants will be discharged from the CRU on Day 6. A follow-up phone call (on CRU visit, if needed), will occur 28-35 days after dosing.

The whole study will last for a minimum of 5 weeks and a maximum of 10 weeks.

ELIGIBILITY:
Inclusion Criteria:

* (HI Cohorts Only): Stable HI that meets criteria for Class A or B of the Child-Pugh classification;
* (all Cohorts): BMI of 17.5 to 38.0 kg/m2

Exclusion Criteria:

* Any condition possibly affecting drug absorption Additional Exclusion Criteria for HI Cohorts Only
* Limited predicted life expectancy
* Hepatic dysfunction secondary to acute ongoing hepatocellular process.
* Signs of clinically active Grade 2, 3 or 4 hepatic encephalopathy.
* Severe ascites and/or pleural effusion
* History of kidney, liver, or heart transplantation.
* Persistent severe, uncontrolled hypertension.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2024-06-27 (Actual); Study Completion 2024-06-27 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of PF-07817883 | Day 1 to Day 6
  Plasma PF-07817883 PK parameters
Area Under the Plasma Concentration-time Profile from Time Zero to Extrapolated Infinite Time (AUCinf) | Day 1 to Day 6
  Plasma PF-07817883 PK parameter
Area Under the Plasma Concentration-time Profile from Time Zero to the Time of the Last Quantifiable Concentration (AUClast) | Day 1 to Day 6
  (Optional) Plasma PF-07817883 parameter

SECONDARY OUTCOMES:
Number of Participants with Non-Serious Adverse Events | Screening to Day 35
  Safety Parameters
Number of Participants with Treatment Emergent Adverse Events | Day 1 to Day 35
  Safety Parameters
Number of Participants with Clinically Significant ECG Abnormalities | Day 1 to Day 6
  ECG parameters include QTcF, QRS, RR interval, PR interval, and Heart Rate
Number of Participants with Clinically Significant Abnormal Vital Signs | Day 1 to Day 6
  Vital Signs parameters include diastolic blood pressure, systolic blood pressure, and pulse rate
Number of Participants with Clinically Significant Abnormal Laboratory Values | Baseline to Day 6
  Blood hematology and Chemistry and Urinalysis
Number of Participants with Serious Adverse Events | Screening to Day 35
  Safety Parameters

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (6):
- United States (6):
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - National Institute of Clinical Research, Garden Grove, California
  - Catalina Research Institute, LLC, Montclair, California
  - Research Centers of America ( Hollywood ), Hollywood, Florida
  - Research Centers of America, Hollywood, Florida
  - Genesis Clinical Research, LLC, Tampa, Florida

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C5091014